CLINICAL TRIAL: NCT07258680
Title: Optimization of the First-line Therapy of T-cell Lymphomas
Brief Title: BrEto-TCL - Defining the Role of Brentuximab and Etoposide for Optimizing First-line Therapy of T-cell Lymphomas
Acronym: BrEto-TCL
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: N.N. Petrov National Medical Research Center of Oncology (Other)
Responsible Party: Principal Investigator, Anastasiia Kolgotina, Oncologist, N.N. Petrov National Medical Research Center of Oncology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BrEto-TCL
Record Dates: First submitted 2025-11-14; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Peripheral T-cell Lymphoma
Keywords: PTCL; Peripheral T-Cell Lymphoma; brentuximab vedotin
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Doxorubicin; Vincristine; Etoposide; Cyclophosphamide; Prednisone; Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 1st group - CHOEP (Active Comparator): Therapy of patients in the 1st group of the study is carried out according to the CHOEP scheme (6 courses with an interval of 21 days)
  Interventions: Drug: Doxorubicin; Drug: Vincristine; Drug: Etoposide; Drug: cyclophosphamide; Drug: Prednisone
- 2nd group - CHOP (Active Comparator): The therapy of patients in the 2nd group of the study is carried out according to the CHOP scheme (6 courses with an interval of 21 days)
  Interventions: Drug: Doxorubicin; Drug: Vincristine; Drug: cyclophosphamide; Drug: Prednisone
- 3rd group - CHP-Bv (Active Comparator): Therapy of patients of the 3rd group of the study is carried out according to the CHP-Bv scheme (6 courses with an interval of 21 days)
  Interventions: Drug: Doxorubicin; Drug: cyclophosphamide; Drug: Prednisone; Drug: Brentuximab Vedotin (Bv)
- 4th group - CHEP-Bv (Active Comparator): The therapy of patients in the 4th group is carried out according to the CHEP-Bv scheme (6 courses with an interval of 21 days)
  Interventions: Drug: Doxorubicin; Drug: Etoposide; Drug: cyclophosphamide; Drug: Prednisone; Drug: Brentuximab Vedotin (Bv)

INTERVENTIONS:
Drug: Doxorubicin — doxorubicin 50 mg/m2, day 1
Drug: Vincristine — vincristine 1.4 mg/m2, (maximum dose 2 mg) day 1
  Arms: 1st group - CHOEP; 2nd group - CHOP
Drug: Etoposide — Etoposide 100 mg/m2, 1-3 days
  Arms: 1st group - CHOEP; 4th group - CHEP-Bv
Drug: cyclophosphamide — cyclophosphamide 750 mg/m2, day 1
Drug: Prednisone — prednisone 100 mg, 1-5 days
Drug: Brentuximab Vedotin (Bv) — brentuximab vedotin 1.8 mg / kg, day 1
  Arms: 3rd group - CHP-Bv; 4th group - CHEP-Bv

SUMMARY:
There is no data comparing the effectiveness of the 4 most relevant first-line therapy programs for peripheral T-cell lymphomas (CHOEP, CHOP, CHEP-BV, CHP-BV) in a single study.

For the first time, the effectiveness and toxicity of various first-line PTCL therapy programs in patients with T-cell lymphoma will be analyzed in the conditions of a single medical center of the N.N.Petrov National Research Medical Center of Oncology and optimal therapeutic tactics will be determined, taking into account significant prognostic factors based on effectiveness and toxicity a specific chemotherapy regimen.

DETAILED DESCRIPTION:
A non-randomized retrospective cohort study with prospective inclusion is planned.

Patients with a confirmed diagnosis of PTCL (who meet the inclusion criteria) who were treated at the same center of the NN Petrov National Medical Cancer Research Center from 2013 to 2024, depending on the first-line therapy regimen, will be included in the retrospective part of the study and divided into 2 groups: Group 1: CHOEP regimen Group 2: CHOP regimen

The prospective part of this study is planned to include patients (who meet the inclusion criteria) who are hospitalized at the NN Petrov National Medical Cancer Research Center for treatment from January 2024 to January 2027. Patients will be divided into 2 groups depending on the chemotherapy regimen:

Group 3: chemoimmunotherapy according to the CHP-BV regimen Group 4: chemoimmunotherapy according to the CHEP-BV regimen Based on the data from the medical documentation of patients, the main statistical indicators of the effectiveness of first-line treatment regimens will be calculated using objective methods for assessing the antitumor effect (PET CT, CT), the toxicity of each of the regimens will be assessed, as well as possible prognostic factors for all patient groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed mature T-cell lymphomas
* absence of acute infectious diseases during treatment diseases, chronic diseases in the stage of decompensation
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2

Exclusion Criteria:

* the presence of a history of other malignant neoplasms during the 5-year period before the start of first-line therapy, In addition to in situ neoplasms treated according to appropriate treatment protocols,
* there are acute infectious diseases and chronic diseases in the decompensation stage.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2013-10 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
complete response rate | Up to 8 months
  - Primary endpoints: the complete response rate - The count of participants with CR per IRF following the completion of study treatment (at end of treatment or at the first assessment after the last dose of study treatment and prior to long-term follow-up) according to the Revised Response Criteria for Malignant Lymphoma.

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 8 months
  Any untoward medical occurrence in a clinical investigational participant administered a medicinal product which does not necessarily have a causal relationship with this treatment.
Progression-free Survival | up to 1 year
  The time from the date of randomization to the date of first documentation of progressive disease (PD), death due to any cause, or receipt of subsequent anticancer chemotherapy to treat residual or progressive disease whichever occurred first.
Overall Survival (OS) | up to 1 year
  The time from randomization to death due to any cause.

IPD SHARING:
Plan to Share IPD: No